CLINICAL TRIAL: NCT00030030
Title: Evaluating Silymarin for Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: R21AT000277-01 (NIH)
Record Dates: First submitted 2002-01-30; First posted 2002-01-31 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Silymarin; milk-thistle extract

INTERVENTIONS:
Drug: Silymarin (milk thistle)

SUMMARY:
To investigate the effect of silymarin, derived from the milk thistle plant, Silybum marianum, in preventing and reversing the complications of chronic infection with hepatitis C virus and/or clearing hepatitis C infections.

DETAILED DESCRIPTION:
The objective of this exploratory project is to assess the feasibility of investigating the effect of silymarin, derived from the milk thistle plant, Silybum marianum, in preventing and reversing the complications of chronic infection with HCV and/or clearing HCV infections, thereby generating preliminary results to serve as the basis of a more definitive study. Allopathic therapeutic interventions have not proved promising, particularly with the genotype most commonly encountered in Egypt and they are prohibitively expensive in the developing world. Egypt has the highest prevalence of HCV infection in the world, averaging 15-25% in rural communities. There are limited rigorous assessments of the dietary supplement milk thistle, but there is promise of salutary effect. The specific aims are to evaluate whether silymarin, the extract of milk thistle, can: (1) improves hepatic morbidity in subjects with chronic HCV hepatitis and/or cirrhosis; (2) prevent progression of liver disease in participants who have chronic HCV infections but who have normal liver enzyme levels; (3) help clear HCV infections; and (4) improves these participants' quality of life. Participants will be randomly assigned to receive silymarin or a vitamin supplement (below antioxidant levels). Participants will be recruited from a cohort of HCV-infected individuals currently enrolled in a large observational study in Egypt. Participants will receive the supplements daily for 18 months, with measures obtained every six months. Measures to be assessed will include: retention in the study, compliance with study assignment, self-described symptoms, alanine aminotransferase (ALT) levels, serum collagen markers, abdominal ultrasound, viral load and clearance, and quality of life (SF36 survey). It is hypothesized that silymarin will not lead to clearance of HCV infections but can prevent progression of liver disease in participants with chronic HCV hepatitis and, in some cases, reverse hepatic lesions that are already present, as well as improving the quality of life in individuals who use this dietary supplement. This exploratory project is anticipated to result in successful initiation of larger and more definitive studies of the effect of milk thistle on HCV infection. Evidence of beneficial effect of an inexpensive and benign herbal dietary supplement would have great impact on the large global population suffering from chronic HCV infection.

Age Groups: Child, Adult, Older Adult
Dates: Start 2000-07; Study Completion 2002-06